CLINICAL TRIAL: NCT05529758
Title: A Third-Wave Intervention for Internalized Weight Bias Combined With a Weight Loss Program Using Video Conferencing Software
Brief Title: Virtual Third-Wave Intervention for Internalized Weight Bias Combined With a Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Caroline Porter-, Graduate Student, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-001438
Record Dates: First submitted 2022-08-19; First posted 2022-09-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Weight Loss; Weight Prejudice
Keywords: Behavioral Weight Loss Program
MeSH Terms: conditions — Weight Loss; Weight Prejudice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Receives internalized weight bias intervention along with standard behavioral weight loss program
  Interventions: Behavioral: Internalized Weight Bias Intervention

INTERVENTIONS:
Behavioral: Internalized Weight Bias Intervention — ACT-based programs and self-compassion have shown promise throughout research for lowering IWB (Berman et al., 2016; Levin et al., 2018; Lillis et al., 2009; Palmeira, Cunha, & Pinto-Gouveia, 2017; Palmeira, Pinto-Gouveia, & Cunha, 2017; Forbes et al., 2020). Therefore, using techniques from prior ACT- and self-compassion based programs, a weight bias reduction intervention will be administered. Session topics will include psychoeducation and coping for weight bias and internal weight bias, and these topics will be viewed through a self-compassionate and ACT-based lens (for example, participants may defuse from internal critical thoughts rather than challenge them). Sessions will also cover acceptance, cognitive defusion, mindfulness, committed action, and the dialectical behavioral therapy (DBT) DEARMAN skill.

SUMMARY:
The current study aims to test a third-wave based IWB intervention paired with a standard BWLP delivered through video conferencing software.

DETAILED DESCRIPTION:
Internalized weight bias (IWB), has been shown to impact mental (e.g., depression and anxiety) and physical health (e.g., cardiometabolic functioning), as well as weight loss and weight loss associated behaviors (e.g., interference with exercise and healthy eating). These associated behaviors especially pose a risk for weight regain and disruption of healthy weight loss. Therefore, given the association between IWB and weight loss associated behaviors, as well as the psychological and health risks associated with IWB, it is clear that IWB interventions are also needed independently and in conjunction with behavioral weight loss programs (BWLPs). Interventions using third-wave strategies (such as acceptance commitment therapy; ACT) have begun to show promise in reducing IWB, but have not yet looked at this therapy in conjunction with a BWLP. Finally, there has also been a growing interest in and need for telehealth-based programs and interventions. The COVID19 pandemic demonstrated a clear need for efficacious telehealth programs, and a further benefit is that these programs may reach populations with limited access to resources (i.e., rural populations). Thus, the current study aims to examine a third-wave based IWB intervention paired with a standard BWLP delivered through video conferencing software.

ELIGIBILITY:
Inclusion:

1. Interested in weight loss
2. 18 or older
3. BMI of 25 kg/m2 or greater
4. Higher-than-average levels of IWB
5. Access to internet, along with a web camera and sound, and be able to use video conferencing software and attend weekly online groups, and access to a reliable scale to weigh themselves weekly

   Exclusion:
6. Individuals with current use of medication prescribed for weight loss (such as orlistat, sibutramine, or rimonabant)
7. Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Weight Change | Baseline to Week 10
  Weight Change
Weight Bias Internalization Scale | Baseline to Week 10
  Internalized Weight Bias, which is internalizing weight bias towards oneself, is scored on a scale of 1 to 7, with higher scores indicating greater weight bias internalization.
Weight Self-Stigma Questionnaire | Baseline to Week 10
  Internalized Weight Bias, which is internalizing weight bias towards oneself, is summed on a scale of 12 to 60, with higher scores indicating greater weight bias internalization. Includes two subscales of Self-Devaluation (WSSQ-SD) and Fear of Enacted Stigma (WSSQ-FNE), each summed on scale of 6-30.
Revised Morgenstern Physical Activity Questionnaire (PAQ-M) | Baseline to Week 10
  The Revised Morgenstern Physical Activity Questionnaire assesses Physical Activity through 11 items, asking participants specifically about light, moderate, or rigorous exercise, recreational activities, home, volunteer, or work activities, and chores.
Diet History Questionnaire III (DHQ III) | Baseline to Week 10
  The Diet History Questionnaire III assesses Eating Behavior, including various food items/groups (with 124 food items) and frequency and portion of each food item or group.
Three Factor Eating Questionnaire-R18 (TFEQ-18) | Baseline to Week 10
  The Three Factor Eating Questionnaire-R18 is an 18-item measure designed to examine eating behavior through three subscales: cognitive restraint, uncontrolled eating and emotional eating using a 4-point Likert scale, using "definitely true" to "definitely false". Higher scores indicate more disordered eating.

SECONDARY OUTCOMES:
Self-Compassion Scale | Baseline to Week 10
  The Self-Compassion Scale is a 12-item scale that uses a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). The scale has six subscales; the first three represent crucial/core components of self-compassion: self-kindness, common humanity, and mindfulness, and the remaining three serve as counters to these core components, with self-judgement, isolation, and overidentification (becoming wrapped up in negative emotions). The three core components are added together, along with reverse-scored counter components, to create an overall score in which higher scores indicate higher self-compassion.
Brief Stigmatizing Situations Inventory | Baseline to Week 10
  The Brief Stigmatizing Situations Inventory is a 10-item scale used to measure experiences of weight stigma, including items such as "Overhearing other people making rude remarks about you in public," on a Likert scale ranging from 0 (never) to 9 (daily), and higher scores indicating more situations encountered.
Depression Anxiety and Stress Scale - 21 Items (DASS-21) | Baseline to Week 10
  The Depression Anxiety and Stress Scale assess depression, stress, anxiety, with score cut off's for...
  * depression: normal: 0-9, mild: 10-12, moderate:13-20, severe: 21-27, and extremely severe: 28-42.
  * anxiety: normal: 0-6, mild: 7-9, moderate: 10-14, severe:15-19, and extremely severe: 20-42.
  * stress: normal: 0-10, mild:11-18, moderate:19-26, severe: 27-34, and extremely severe: 35-42.
  Higher scores equate higher depression, anxiety, and stress.
Rosenberg Self-Esteem Scale | Baseline to Week 10
  Self-Esteem will be measured utilizing the 10-item Rosenberg Self-Esteem Scale (RSES). The RSES uses a 4-point Likert scale from 1 (strongly disagree) to 4 (strongly agree), which higher scores indicating higher self-esteem.
The Acceptance and Action Questionnaire - Second Edition (AAQ-II) | Baseline to Week 10
  The Acceptance and Action Questionnaire is a 7-item questionnaire that uses a 7-point Likert scale from 1 (never true) to 7 (always true). Higher scores indicate less psychological flexibility and higher experiential avoidance.
Satisfaction with Therapist and Therapy Scale | Baseline to Week 10
  The Satisfaction with Therapist and Therapy Scale assesses satisfaction with therapy and therapist using a 5-point Likert scale, from 1 (Strongly Disagree) to 5 (Strongly Agree). Questions regarding treatment will be adapted for the telehealth, BWLP situation (i.e., "I am satisfied with the quality of the therapy I received" will be adapted to "I am satisfied with the quality of the telehealth weight loss treatment I received"). Similarly, questions about the therapist will be changed to "weight loss coach."
Ruminative Response Scale - Short Form | Baseline to Week 10
  The Ruminative Response Scale - Short Form includes nine items with two subscales; brooding and reflection. The form utilizes a 4-point Likert scale ranging from 1 ("almost never") to 4 ("almost always") for various aspects of rumination. Higher scores indicate more rumination.
Universal Measure of Bias (UMB-FAT) | Baseline to Week 10
  The Universal Measure of Bias (UMB-FAT) is a 20-item scale that assesses attitudes towards fat, using a 7-point scale with "strongly agree" to "strongly disagree." It includes four subscales: negative judgment (dislike towards individuals with overweight or obesity), distance (comfort with individuals with overweight or obesity in social situations), equal rights (assessing the belief that individuals with overweight or obesity deserve legal protection against discrimination) and attraction (the extent to which the participant finds individuals with overweight or obesity to be attractive). Higher scores indicating greater weight bias by the participant.
The Eating Disorder Diagnostic Scale | Baseline to Week 10
  The Eating Disorder Diagnostic Scale - DSM 5 Version is 22-item a questionnaire designed to assess symptoms of anorexia nervosa, bulimia nervosa, and binge-eating disorder per DSM-5 criteria. The questions vary in terms of format, using 6-point Likert ratings from "Not at all" to "Extremely," dichotomous items and asking about frequency of diagnostically relevant behavior over a set period of time (i.e., days per week for over X amount of months)

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Miller, MA, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be kept confidential.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT05529758/Prot_SAP_ICF_000.pdf